CLINICAL TRIAL: NCT00644397
Title: Plate Fixation of Distal Femur Fractures: a Protocol for a Randomized, Prospective Study of Two Plate Options
Brief Title: Plate Fixation of Distal Femur Fractures: A Protocol for a Study of Two Plate Options
Status: Completed | Type: Observational
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Heather A. Vallier, Professor of Orthopaedic Surgery, MetroHealth Medical Center
Other Study IDs: IRB06-00029
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Femoral Fractures
Keywords: distal femur fracture; locked plates; functional outcomes; cost management; femur head; femur neck
MeSH Terms: conditions — Femoral Fractures; Femoral Fractures, Distal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Blade Plate Group: 95-degree Angled Blade Plate
  Interventions: Device: 95-degree Angled Blade Plate
- Locking Plate Group: 4.5mm Condylar Locking Plate
  Interventions: Device: 4.5mm Condylar Locking Plate

INTERVENTIONS:
Device: 95-degree Angled Blade Plate
  Groups: Blade Plate Group
Device: 4.5mm Condylar Locking Plate
  Groups: Locking Plate Group

SUMMARY:
Internal fixation of femur fractures improves alignment and provides stability to the bone and the surrounding soft tissues. This generally allows for early motion of the adjacent joints; thus maximizing overall function of the limb. Open reduction and internal fixation with plates and screws is the standard method that has been used in the treatment of distal femoral fractures. One common traditional method of internal fixation is the 95-degree angled blade plate. Recent advances in technology for distal femur fractures include the LCP™ Condylar Plate. This implant differs from the blade plate, because the LCP offers multiple points of fixed angle contact between the plate and screws in the distal femur. The introduction of plates with the option of locked screws has provided means to increase the rigidity of fixation in osteoporotic bone or in periarticular fractures with a small distal segment, and the LCP may be technically easier to apply than the blade plate. To the investigators' knowledge, there have been no published clinical or biomechanical studies specific to the LCP Condylar Plate, although the early results of LCP implants for other fractures are promising. The investigators believe that locked plating represents a valuable advancement in fracture treatment. However, the limitations of this new technology and the indications for its use have not been completely elucidated. Furthermore, the cost of the new technology is approximately seven times more than the traditional treatment. This is a randomized, prospective, multi-center study to compare the blade plate and the LCP in the distal femur. All patients 16 years of age or older, regardless of race or gender, with a supracondylar fracture of distal femur will be considered. Whether patients are treated with a blade plate or/and LCP, they will be receiving standard orthopedic care for their injury. Neither of these methods currently places a patient at increased surgical or post-surgical risk for problems with infection, nonunion, malunion, or other complications. Because of the study, early and late complication rates and functional outcomes after these treatments may be better defined, allowing for optimization of care of people with these injuries in the future. This should reduce not only direct and indirect costs to the individual, but also costs to society.

ELIGIBILITY:
Inclusion Criteria:

* Closed or Gustilo 13,14 Type I, II or IIIA open fractures that can be treated with an angled blade plate or an LCP Condylar Plate (Orthopaedic Trauma Association fracture classification 33-A, 33- C1, 33- C2), (Tables 1 & Figure 3)
* 16 or more years of age and skeletally-mature, regardless of race or gender

Exclusion Criteria:

* Pathologic fractures secondary to neoplasm
* Time elapsed since injury greater than 10 days before fixation
* Open fractures unable to undergo debridement and irrigation in the first 24 hours
* Inability or refusal to give consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participating research centers will evaluate for enrollment all patients presenting with distal femur fractures. The number of patients to be recruited is based on previously reported malunion rates. Assuming a 15% incidence of malunion in the locked plating group, a difference of +/- 5% would be statistically significant. In order for the study to have power of 80% to detect a difference at the 0.05 level, 49 patients will be required in each group.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2006-05; Primary Completion 2018-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather A. Vallier, M.D., Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Claireaux HA, Searle HKC, Parsons NR, Griffin XL. Interventions for treating fractures of the distal femur in adults. Cochrane Database Syst Rev. 2022 Oct 5;10(10):CD010606. doi: 10.1002/14651858.CD010606.pub3. PMID 36197809